CLINICAL TRIAL: NCT06675084
Title: Mortality and Rehospitalization Risk Assessment by Skilled Caregivers Compared to Existing Tools in Acute Geriatric Departments
Status: Not yet recruiting | Type: Observational
Sponsor: Shmuel Harofeh Hospital, Geriatric Medical Center (Other Government)
Responsible Party: Principal Investigator, Yochai Levy, Hospital deputy director, Shmuel Harofeh Hospital, Geriatric Medical Center
Other Study IDs: SH-120-24
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Clinical Decision Support
Keywords: Geriatric, acute care, older adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mortality and Rehospitalization Risk Assessment by Skilled Caregivers Compared to Existing Tools in Acute Geriatric Departments

Background The elderly population in Israel and worldwide is steadily increasing, leading to greater demand for medical services, including palliative care. In 2019, individuals aged 65+ accounted for 64% of hospital admissions and 70% of hospital days in Israel. Approximately 19% of these were readmissions, a rate that increases with age. Effective tools for identifying patients at high risk of rehospitalization and mortality are lacking, which, if improved, could benefit patients through targeted palliative and end-of-life care. Enhanced tools could reduce unnecessary interventions, improve patient well-being, and alleviate economic burdens on healthcare.

Research Objectives

1. Evaluate mortality and rehospitalization rates in acute geriatric departments.
2. Identify risk factors for rehospitalization and mortality in acutely hospitalized elderly patients.
3. Compare the effectiveness of skilled caregiver assessments versus validated prediction tools for mortality and rehospitalization within one year.

Hypotheses

1. Mortality and rehospitalization rates in acute geriatric departments are comparable to those in internal medicine.
2. Multiple factors-such as age, family support, comorbidities, functional and cognitive status-correlate with mortality risk.
3. Skilled caregiver assessments predict mortality and rehospitalization more accurately than existing validated tools.

Study Design Type: Prospective cohort observational study. Location: Shmuel Harofe Hospital.

Study Population Participants are elderly patients admitted to acute geriatric departments at Shmuel Harofe Hospital for acute conditions. Approximately 600 participants will be recruited, with an additional 200-300 if statistical analysis reveals trends.

Recruitment Period: Two years. Follow-up Period: Up to one year post-admission.

Methods and Materials

Data will be collected on demographic, functional, cognitive, and emotional factors, as well as clinical history, hospital admissions, comorbidities, and lab results. Predictive assessments will include:

1. Mortality Prediction using the WALTER Index for the elderly.
2. Rehospitalization Risk using the LACE Index, validated for 30-day readmission risk.
3. Subjective Caregiver Assessments from geriatric specialists and nursing supervisors, estimating life expectancy and 30-day, 3-month, and 1-year rehospitalization risk.

Data Analysis Data will be coded and statistically analyzed without interventions outside of standard care. The WALTER and LACE indices will utilize existing clinical data.

Ethical Considerations As this is an observational study without intervention, a waiver for informed consent was granted.

Importance of Research Early identification of high-risk patients will enable preventive interventions, support transitions to palliative care where appropriate, and promote advance directives, ultimately improving patient care and reducing healthcare costs by preventing costly, unnecessary readmissions and interventions.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to acute geriatric departments at Shmuel Harofe Hospital for acute conditions.

-

Exclusion Criteria: 1. Admission for social reasons. 2. Patients under palliative end of life care.

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old admitted to acute geriatric departments at Shmuel Harofe Hospital for acute conditions.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness of skilled caregiver assessments versus validated prediction tools for mortality and rehospitalization within one year | 2 years

SECONDARY OUTCOMES:
Identify risk factors for rehospitalization and mortality in acutely hospitalized elderly patients. | 2 years

IPD SHARING:
Plan to Share IPD: No